CLINICAL TRIAL: NCT00340938
Title: Family Management of Childhood Diabetes Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999905030; 05-CH-N030
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2019-11-01

CONDITIONS: Diabetes; Type 1 Diabetes
Keywords: Adherence; Education; Problem Solving; Motivation; Locus of Responsibility
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Hematologic Tests

INTERVENTIONS:
Procedure: Blood testing

SUMMARY:
This study will test the effectiveness of a practical, low-cost, problem-solving method called WE CAN that can be taught to families at diabetes clinics. The goal is to see if this teaching and support can help with controlling the level of blood sugar in children with type 1 diabetes as they approach adolescence. Attention would go to young people's completion of tasks necessary to manage diabetes, quality of life, and psychological adjustments, plus the role of the family in these situations. Type 1 diabetes mellitus, accounting for less than 10% of the disease cases, is marked by the inability of the pancreas to secrete insulin. People who have it must consistently manage their disease. Successful disease management for children depends on the family's adaptation to treatment demands. Yet maintaining acceptable blood sugar control becomes more difficult for adolescents, owing to changes in the body during that period of life. Also, early adolescence is a vital time in people's development of health outcomes. The title WE CAN is a way to remember the steps of the problem-solving method:

* Work together to set goals
* Explore barriers and solutions
* Choose the best solutions
* Act on your plan
* Note the results

Children who have reached age 9 but are not yet 14.5 years who have had type 1 diabetes for at least 1 year and who have had at least two visits to diabetes clinics at one of four clinical sites may be eligible for this study. A total of 120 children will participate in clinic visits once every 3 months.

Participants and their families will attend diabetes clinic visits once every 3 months. They will be assigned to one of two groups: standard care or WE CAN. Those in the WE CAN group will have visits about 15 to 45 minutes longer than those involved in the standard care group. All participants will have two home visits: at the beginning and at 6 months. There will also be telephone interviews, about 20 minutes long, once every 3 months with the children and their parents. Medical data will be collected during each visit to the clinic, including blood samples. A health advisor will work with the families. Questionnaires given to parents and children separately will measure diabetes-related family conflict, parent child sharing of responsibilities for the disease, attitudes and emotions about diabetes, and impact of the disease on the child's life. Also, parents and children together will take part in a 10-minute discussion of a diabetes-related issue that has caused friction among family members. They will discuss the problem, come up with possible solutions, and to try to decide on a solution within 10 minutes. Family discussions will be videotaped at the first home visit and at the 6-month home visit.

Families in both groups will receive more detailed monitoring of family diabetes management than is usually the case. Those in the WE CAN group may be able to control diabetes more effectively during the child's early adolescence, though that result is not guaranteed. If the family guidance and support provided by the WE CAN health advisor is effective, children in that group may have better results in blood sugar than they would if they did not participate in the study. Each family member completing the first and 6-month visits and completing each telephone interview will receive payment for participating.

DETAILED DESCRIPTION:
This protocol describes a multi-center, randomized controlled trial to test whether a clinic-integrated, low intensity, multi-component behavioral intervention is effective in preventing the deterioration in glycemic control, treatment adherence, and quality of life that commonly occur during late childhood and early adolescence in youth with type 1 diabetes. The study will also examine mechanisms and processes that influence the effectiveness of family management of diabetes during this developmental period.

ELIGIBILITY:
* INCLUSION CRITERIA - CHILD CRITERIA:

Age 9.0 to 14.5

Type I diabetes diagnosis (diagnosed by ADA criteria) for a minimum of 1 year requiring insulin treatment

Insulin dose greater than or equal to 0.5 u/kg/day

Mean A1c over last 8 months is less than 13.0%

No major chronic diseases (except well-controlled thyroid, asthma)

No major visual/auditory impairments

Child is not in self-contained special education class throughout the school day

No DSM-IV diagnosis of bipolar, addiction, psychosis, or eating disorder documented in existing medical chart. No record of inpatient hospitalization for mental disorder in past six months including substance abuse rehabilitation, eating disorder units or day treatment programs. No history of anti-psychotic medications for the past 6 months.

No diagnosis of mental retardation.

Literate (reading, writing) in English/Spanish at 2nd grade level

Willing to provide informed assent

Children who are currently enrolled in any other study (observational or interventional) are not eligible for enrollment. Children cannot enroll in another study during the course of this study. Those who have been in an intervention arm of a trial of a behavioral, psychological or psychoeducational intervention and concluded their study follow-up within the past 12 months are also ineligible to participate. However, children who were in a standard care control group in an intervention study or who were in an observational study are eligible once they have completed all scheduled study follow-ups.

PARENT/FAMILY ENVIRONMENT CRITERIA:

Child lives in geographically stable home, no multiple foster homes, boarding school, or institutions expected to next 2 years.

The same 1 or 2 adult caregivers have accompanied the child to every diabetes clinic visit in the past year, and a single adult, who has primary responsibility for the child's diabetes care and monitoring, agrees to participate in all aspects of the protocol (single-parent families, blended families and separated parents will be eligible).

Family has no plan to re-locate out of area within the next 2 years of the study.

Home has telephone access

Primary parent is not currently undergoing treatment for substance abuse.

Primary parent has not been hospitalized in past 6 months for mental disorder.

Primary caretaker has no history of psychosis.

Child had at least 2 clinic visits within last 12 months

Parent and child wiling to come to clinic every 3 months for duration (2 years) of study.

Families who are currently enrolled in any other study (observational or interventional) are not eligible for enrollment. Families cannot enroll in another study during the course of this study. Those who have been in an intervention arm of a trial of a behavioral, psychological or psychoeducational intervention and concluded their study follow-up within the past 12 month are also ineligible to participate. However, families who were in a standard care control group in an intervention study or who were in an observational study are eligible once they have completed all scheduled study follow-ups.

If a family has more than one eligible child, all qualifying children who provide consent/assent will participate in assessment and intervention or control activities; however, only the oldest qualifying child will be included in statistical analyses.

Ages: 9 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1298 (Actual)
Dates: Start 2004-11-08; Primary Completion 2009-03-01 (Actual); Study Completion 2009-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonja R. Nansel, Ph.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (3):
- United States (3):
  - Childrens Memorial Hospital, Chicago, Chicago, Illinois
  - Joslin Diabetes Center, Boston, Massachusetts
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Background] Allen DA, Tennen H, McGrade BJ, Affleck G, Ratzan S. Parent and child perceptions of the management of juvenile diabetes. J Pediatr Psychol. 1983 Jun;8(2):129-41. doi: 10.1093/jpepsy/8.2.129. No abstract available. PMID 6875761
- [Background] Amiel SA, Sherwin RS, Simonson DC, Lauritano AA, Tamborlane WV. Impaired insulin action in puberty. A contributing factor to poor glycemic control in adolescents with diabetes. N Engl J Med. 1986 Jul 24;315(4):215-9. doi: 10.1056/NEJM198607243150402. PMID 3523245
- [Background] Anderson BJ, Brackett J, Ho J, Laffel LM. An office-based intervention to maintain parent-adolescent teamwork in diabetes management. Impact on parent involvement, family conflict, and subsequent glycemic control. Diabetes Care. 1999 May;22(5):713-21. doi: 10.2337/diacare.22.5.713. PMID 10332671